CLINICAL TRIAL: NCT01192360
Title: Dynamic Contrast Enhanced Magnetic Resonance Perfusion Imaging in Congenital Heart Disease and Lung Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Lars Grosse-Wortmann, Principal Investigator, The Hospital for Sick Children
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1000016503
Record Dates: First submitted 2010-08-30; First posted 2010-09-01 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Heart Disease; Cystic Fibrosis; Asthma
Keywords: pediatrics; Heart Disease; Cystic Fibrosis; Severe Asthma; Magnetic Resonance Imaging
MeSH Terms: conditions — Heart Diseases; Cystic Fibrosis; Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cardiac Patients (Experimental): In addition to the routine clinical MRI, we will conduct the DCE MR perfusion imaging research component. For this, we will measure native pre-contrast T1 and then inject a tight bolus of gadolinium (0.1mmol/kg) while acquiring high temporal resolution T1-weighted 3D contrast dynamics information over the whole thorax while the patient is holding his / her breath. Overall, the research component will prolong the clinical study by approximately 5 minutes.
  Interventions: Procedure: Phase contrast flow velocity mapping (PC); Procedure: Dynamic contrast-enhanced magnetic resonance imaging
- Pulmonary Patients (Experimental): Patients in this group will receive a full cardiac and pulmonary MRI assessment, with the DCE pulmonary perfusion scan added as described above. Overall, the investigation will take approximately 45 minutes
  Interventions: Procedure: Phase contrast flow velocity mapping (PC); Procedure: Dynamic contrast-enhanced magnetic resonance imaging

INTERVENTIONS:
Procedure: Phase contrast flow velocity mapping (PC) — An MRI is done using the phase contrast flow velocity mapping (PC)technique. Using PC, an imaging slice is prescribed perpendicular to the vessel's course. Within the pulmonary circulation, PC can quantify total pulmonary blood flow and the right / left distribution of the lung blood flow volume.
Procedure: Dynamic contrast-enhanced magnetic resonance imaging — Dynamic contrast-enhanced magnetic resonance (DCE MR) perfusion imaging imaging is a non-invasive method to quantify regional pulmonary blood flow. A bolus of gadolinium-containing contrast medium is injected and its passage through the pulmonary circulation traced using a repetitive rapid three-dimensional (3D) T1 weighted angiography sequence.

SUMMARY:
The primary objective of this study is to determine if quantitative Dynamic contrast-enhanced magnetic resonance (DCE MR) perfusion imaging accurately quantifies right and left pulmonary artery blood flow as compared with phase contrast flow velocity mapping (PC), the current gold standard of flow volume measurements.

DETAILED DESCRIPTION:
Many conditions of the heart or the lungs lead to differences in how the blood is pumped to the lungs. Specifically, some areas of the lung may receive less blood supply than others. We would like to do a research study in children and adolescents who have a heart condition or a chronic or stable lung condition. We are doing this study to see if measuring the circulation of blood in the lungs in children is possible using magnetic resonance imaging (MRI) with a special dye (contrast medium) injection called Magnevist®.

ELIGIBILITY:
Inclusion Criteria:

Cardiac Patients:

1. Patients > 6 years of age
2. Patients with suspected or confirmed congenital or acquired heart disease
3. Who undergo a clinically indicated MRI scan, including gadolinium (MRI contrast medium)
4. And receive gadolinium (= MRI contrast medium) as part of their clinical investigation

Pulmonary Patients:

1. Patients > 6 years of age
2. Patients with a chronic and stable lung condition, such as cystic fibrosis, severe asthma.

Exclusion Criteria:

1. Children under the age of 6 will be excluded as they are routinely scanned under general anesthesia
2. Patients in whom MRI is contraindicated (e.g. pacemaker, ocular metal, claustrophobia, tattoos)
3. Patients with a known allergy to gadolinium.
4. Patients with a history of allergic disposition or have anaphylactic reactions
5. Moderate-to-severe renal impairment (defined as having a GFR/ eGFR < 60 mL/min)
6. Have Sickle Cell anemia
7. Known pregnancy, or breast feeding
8. Patient is uncooperative during a MRI without sedation or anesthesia

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Pulmonary blood flow | 1 hour
  Pulmonary blood flow as measured with DCE MRI perfusion imaging will be compared to MRI phase contrast imaging, which is the gold standard of non-invasive flow measurements.

SECONDARY OUTCOMES:
Perfusion defects detected | 1 hour
  Perfusion defects (number and location) will be compared to images of lung morphology and correlated with pathology within the lung parenchyma and central airways.
Quantitative results from dynamic contrast-enhanced magnetic resonance perfusion imaging | 1 hour
  Quantitative results from DCE MRI perfusion imaging (including mean transit time, pulmonary blood flow, pulmonary blood volume) will be correlated with the results of pulmonary perfusion tests, where clinically available.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Grosse-Wortmann, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada